CLINICAL TRIAL: NCT01403064
Title: A Phase 2, Multi-center, Randomized, Double-blind, Placebo-controlled Clinical Trial to Evaluate the Safety and Efficacy of ALD518 in the Reduction of Oral Mucositis in Subjects With Head and Neck Cancer Receiving Concomitant Chemotherapy and Radiotherapy
Brief Title: Safety and Efficacy of ALD518 for Reducing Oral Mucositis in Head and Neck Cancer Subjects
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: due to lack of efficacy
Sponsor: CSL Behring (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ALD518-CLIN-009
Record Dates: First submitted 2011-07-25; First posted 2011-07-27 (Estimated); Results first posted 2021-05-11 (Actual); Last update posted 2021-05-11 (Actual); Status verified 2021-04

CONDITIONS: Oral Mucositis
Keywords: Oral mucositis; head and neck cancer; chemotherapy; radiotherapy
MeSH Terms: conditions — Stomatitis; Head and Neck Neoplasms | interventions — clazakizumab; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Open Label ALD518 (Experimental)
  Interventions: Biological: ALD518
- ALD518 Dose 1 (Experimental)
  Interventions: Biological: ALD518
- ALD518 Dose 2 (Experimental)
  Interventions: Biological: ALD518
- Placebo (Placebo Comparator)
  Interventions: Drug: 0.9% saline

INTERVENTIONS:
Biological: ALD518 — IV
  Arms: ALD518 Dose 1; ALD518 Dose 2; Open Label ALD518
Drug: 0.9% saline — IV Infusion
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of ALD518 in modifying the course of oral mucositis in subjects with head and neck cancer receiving concomitant chemotherapy and radiotherapy

DETAILED DESCRIPTION:
This was a Phase 2, placebo-controlled, double-blind study in subjects newly diagnosed with head and neck cancer (who had not received previous treatment for oral mucositis) and who were receiving concomitant chemotherapy and radiotherapy. Subject eligibility, including tumor staging, was assessed during the screening period, which was to occur within 30 days prior to the initiation of radiation therapy. The radiation therapy treatment period was approximately 7 weeks, depending on the subject's prescribed radiation plan. Prior to the randomized portion of the trial, the first 7 subjects enrolled in the study entered a safety run-in evaluation and received a total of 2 doses of open-label clazakizumab 160 mg IV, 4 weeks apart (Day 0 and Week 4 of radiation); these subjects were not eligible for the randomized portion of the study. Subsequent to completion of the safety run-in, eligible subjects were randomized 1:1:1 to treatment with 2 doses of clazakizumab 160 mg, or clazakizumab 320 mg, or placebo, administered IV 3 weeks apart (Day 0 and Week 3 of radiation therapy). All subjects were to be followed for 4 weeks post last day of radiotherapy treatment for the primary efficacy and safety assessments and then for up to an additional 12 months of long-term follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Have recently diagnosed (< than 6 months prior to screening visit date), pathologically confirmed, non-metastatic SCC of the oral cavity, oropharynx, hypopharynx or larynx that will be treated with CRT as first-line treatment; subjects with a history of surgical management (approximately 4-6 weeks before RT with sufficient time for post-surgical healing) are eligible
* Have a plan to receive a continuous course of conventional external beam irradiation delivered by intensity-modulated radiotherapy (IMRT) as single daily fractions of 2.0 to 2.2 Gy, with a cumulative radiation dose between 55 and 72 Gy.
* Have a plan to receive a standard cisplatin CT regimen administered tri-weekly (80 to 100 mg/m2, on Days 0, 21, and 42) or weekly (30 to 40 mg/m2) or a standard carboplatin regimen administered weekly (100 mg/m2)
* Have an Eastern Cooperative Oncology Group (ECOG) performance status ≤ 1
* CRP < 80 mg/L
* Have adequate hematopoietic, hepatic, and renal function at the screening visit

Exclusion Criteria:

* Tumor of the lips, sinuses, salivary glands, nasopharynx or unknown primary tumor
* Metastatic disease (M1) Stage IV C
* Any prior history of head and neck cancer
* Prior radiation to the head and neck
* Have had a major surgical procedure, other than for HNC, or significant traumatic injury within 4 weeks prior to the initiation of RT; or anticipation of need for a major surgical procedure during the clinical trial
* Active infectious disease, excluding oral candidiasis
* Have OM at the screening visit
* Have a history of hypersensitivity to monoclonal antibody

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Actual)
Dates: Start 2011-07; Primary Completion 2013-04 (Actual); Study Completion 2014-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey Smith, MD FRCP, Study Director — Alder Biopharmaceuticals, Inc.
Locations (31):
- United States (13):
  - Morton Plant Mease Health Care, Clearwater, Florida
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Karmanos Cancer Center, Detroit, Michigan
  - Detroit Clinical Research Center, Farmington Hills, Michigan
  - John Theurer Cancer Center at Hackensack University Medical Center, Hackensack, New Jersey
  - University of New Mexico Cancer Center, Albuquerque, New Mexico
  - Mount Sinai School of Medicine, New York, New York
  - SUNY Upstate Medical University, Syracuse, New York
  - Temple University Hospital, Philadelphia, Pennsylvania
  - Spartanburg Regional Medical Center, Spartanburg, South Carolina
  - Cancer Specialists of Southern Texas, Corpus Christi, Texas
  - University of Texas Southwestern Medical Center, Dallas, Texas
  - VA Puget Sound Health Care Syatem, Seattle, Washington
- Australia (6):
  - St. Vincent's Hospital, Darlinghurst, New South Wales
  - Calvary Mater Newcastle, Waratah, New South Wales
  - Royale Brisbane and Women's Hospital, Herston, Queensland
  - Princess Alexandra Hospital, Woolloongabba, Queensland
  - Adelaide Radiotherapy Centre, Adelaide, South Australia
  - Royal Adelaide Hospital, Adelaide, South Australia
- Austria (3):
  - LKH Graz, HNO Ambulanz, Graz
  - Univ. Klinik fur Innere Medizin III, Salzburg
  - Hanusch Krankenhaus, Vienna
- Canada (3):
  - Cancer Centre of Southeastern Ontario, Kingston, Ontario
  - Maisonneuve-Rosemont Hospital, Montreal, Quebec
  - CHUQ-L'Hotel-Dieu de Quebec, Québec
- Germany (3):
  - Uniklinik Koln, Cologne
  - Universitatsklinikum Freiburg, Freiburg im Breisgau
  - University Medical School, Saarland, Homburg
- Italy (3):
  - A.O. San Paolo - Polo Universitario, Milan
  - Istituto Nazionale dei tumari, Milan
  - Azienda Ospedaliero-Universitaria Santa Maria della Misericordia, Udine

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: 0.9% saline administered as two intravenous infusions (IV) 3 weeks apart
- ALD518 (160 mg, OL): ALD518 160 mg IV every 4 weeks for a total of 2 doses in open-label (OL) treatment
- ALD518 (160 mg, R): ALD518 160 mg IV every 3 weeks for a total of 2 doses in randomized (R) treatment
- ALD518 (320 mg, R): ALD518 320 mg IV every 3 weeks for a total of 2 doses in randomized (R) treatment
Period: Overall Study
Arm/Group | Placebo | ALD518 (160 mg, OL) | ALD518 (160 mg, R) | ALD518 (320 mg, R)
Started | 24 | 7 | 23 | 22
Completed | 23 | 7 | 19 | 19
Not Completed | 1 | 0 | 4 | 3
Not completed — Death | 0 | 0 | 1 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 1 | 1
Not completed — Other | 1 | 0 | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | ALD518 (160 mg, OL) | ALD518 (160 mg, R) | ALD518 (320 mg, R) | Total
Number analyzed (Participants) | 24 | 7 | 23 | 22 | 76
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.8 (7.92) | 56.3 (11.93) | 58.6 (7.43) | 55.1 (7.18) | 57.4 (8.00)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 1 | 7 | 1 | 13
  Male | 20 | 6 | 16 | 21 | 63
Region of Enrollment [Number; unit: participants]
  Canada | 0 | 0 | 0 | 1 | 1
  Austria | 0 | 0 | 1 | 4 | 5
  United States | 7 | 6 | 5 | 8 | 26
  Italy | 3 | 0 | 5 | 4 | 12
  Australia | 9 | 1 | 2 | 3 | 15
  Germany | 5 | 0 | 10 | 2 | 17

OUTCOME MEASURES:

1. Primary Outcome: Percent of Participants With Adverse Events, Serious Adverse Events and Clinically Significant Laboratory Abnormalities
Time Frame: Up to 15 months
Population: Safety Population (SP) defined as any subject who received at least 1 dose of ALD518 or placebo. Subjects were analyzed based on the treatments they received. As pre-specified, the two treatment groups that received 160 mg (open label and randomized) were combined into one 160 mg group for analysis purposes of this endpoint.
Measure: Number; unit: percentage of participants
Groups:
- ALD518 (160 mg): ALD518 160 mg IV every 4 weeks for a total of 2 doses in open-label (OL) treatment or ALD518 160 mg IV every 3 weeks for a total of 2 doses in randomized (R) treatment
- ALD518 (320 mg): ALD518 320 mg IV every 3 weeks for a total of 2 doses in randomized (R) treatment
Arm/Group | Placebo | ALD518 (160 mg) | ALD518 (320 mg)
Number analyzed (Participants) | 23 | 32 | 21
percentage of participants
  Adverse events (AEs) | 95.7 | 100 | 100
  Serious adverse events | 30.4 | 46.9 | 38.1
  Clinically significant laboratory abnormalities | 0 | 6.3 | 4.8
  Treatment-related AEs | 52.2 | 65.6 | 57.1
  AEs leading to treatment discontinuation | 0 | 3.1 | 4.8

2. Primary Outcome: Number of Participants With Adverse Events, Serious Adverse Events and Clinically Significant Laboratory Abnormalities
Time Frame: Up to 15 months
Population: SP. As pre-specified, the two treatment groups that received 160 mg (open label and randomized) were combined into one 160 mg group for analysis purposes of this endpoint.
Measure: Number; unit: participants
Arm/Group | Placebo | ALD518 (160 mg) | ALD518 (320 mg)
Number analyzed (Participants) | 23 | 32 | 21
participants
  Adverse events (AEs) | 22 | 32 | 21
  Serious adverse events | 7 | 15 | 8
  Clinically significant laboratory abnormalities | 0 | 2 | 1
  Treatment-related AEs | 12 | 21 | 12
  AEs leading to treatment discontinuation | 0 | 1 | 1

3. Primary Outcome: Percent of Participants With All Grades of Oral Mucositis (OM) at a Radiation Dose of 55 Gy
Description: Gray (Gy) is used as a unit of the radiation quantity absorbed dose that measures the energy deposited by ionizing radiation in a unit mass of matter being irradiated, and is used for measuring the delivered dose of ionizing radiation in applications such as radiotherapy. The 55 Gy ulcerative OM assessment is defined as the first ulcerative OM assessment that occurred on the day of or after the subject received the radiation therapy that first resulted in their cumulative dose of radiation being ≥ 55 Gy
Time Frame: Up to 12 weeks
Population: Full Analysis Population (FAP) defined as those randomized subjects who received at least 1 dose of ALD518 or placebo. Subjects were analyzed based on the treatments to which they were assigned.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | ALD518 (160 mg, OL) | ALD518 (160 mg, R) | ALD518 (320 mg, R)
Number analyzed (Participants) | 24 | 7 | 23 | 22
percentage of participants | 79.2 | 71.4 | 100 | 77.3

4. Primary Outcome: Number of Participants With All Grades of OM at a Radiation Dose of 55 Gy
Description: The 55 Gy ulcerative OM assessment is defined as the first ulcerative OM assessment that occurred on the day of or after the subject received the radiation therapy that first resulted in their cumulative dose of radiation being ≥ 55 Gy
Time Frame: Up to 12 weeks
Population: FAP
Measure: Number; unit: participants
Arm/Group | Placebo | ALD518 (160 mg, OL) | ALD518 (160 mg, R) | ALD518 (320 mg, R)
Number analyzed (Participants) | 24 | 7 | 23 | 22
participants | 19 | 5 | 23 | 17

5. Secondary Outcome: Percent of Participants With Ulcerative OM at Varying Cumulative Radiation Doses (Gy)
Description: The ulcerative OM assessment at a specific cumulative radiation dose (35 Gy, 45 Gy, 55 Gy or 65 Gy) is defined as the first ulcerative OM assessment that occurred on the day of or after the subject received the radiation therapy that first resulted in the specific cumulative dose of radiation being ≥35 Gy, ≥45 Gy, ≥55 Gy or≥ 65 Gy
Time Frame: Up to 12 weeks
Population: FAP, 3 participants missing data
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | ALD518 (160 mg, OL) | ALD518 (160 mg, R) | ALD518 (320 mg, R)
Number analyzed (Participants) | 24 | 7 | 22 | 20
percentage of participants
  35 Gy | 58.3 | 85.7 | 81.8 | 65.0
  45 Gy | 87.5 | 85.7 | 90.9 | 75.0
  55 Gy | 79.2 | 71.4 | 100 | 75.0
  65 Gy: number analyzed (Participants) | 18 | 6 | 19 | 16
  65 Gy | 83.3 | 83.3 | 100 | 68.8

6. Secondary Outcome: Number of Participants With Ulcerative OM at Varying Cumulative Radiation Doses (Gy)
Description: as for outcome 5
Time Frame: Up to 12 weeks
Population: FAP, 3 participants missing data
Measure: Number; unit: participants
Arm/Group | Placebo | ALD518 (160 mg, OL) | ALD518 (160 mg, R) | ALD518 (320 mg, R)
Number analyzed (Participants) | 24 | 7 | 22 | 20
participants
  35 Gy | 14 | 6 | 18 | 13
  45 Gy | 21 | 6 | 20 | 15
  55 Gy | 19 | 5 | 22 | 15
  65 Gy: number analyzed (Participants) | 18 | 6 | 19 | 16
  65 Gy | 15 | 5 | 19 | 11

7. Secondary Outcome: Percent of Participants With Severe OM at Varying Cumulative Radiation Doses (Gy)
Description: The severe OM assessment at a specific cumulative radiation dose (35 Gy, 45 Gy, 55 Gy or 65 Gy) is defined as the first severe OM assessment that occurred on the day of or after the subject received the radiation therapy that first resulted in the specific cumulative dose of radiation being ≥35 Gy, ≥45 Gy, ≥55 Gy or≥ 65 Gy
Time Frame: Measured from onset of OM through Week 12
Population: FAP, 3 participants missing data
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | ALD518 (160 mg, OL) | ALD518 (160 mg, R) | ALD518 (320 mg, R)
Number analyzed (Participants) | 24 | 7 | 22 | 20
percentage of participants
  35 Gy | 25.0 | 57.1 | 27.3 | 30.0
  45 Gy | 41.7 | 71.4 | 36.4 | 45.0
  55 Gy | 50.0 | 71.4 | 40.9 | 55.0
  65 Gy: number analyzed (Participants) | 18 | 6 | 19 | 16
  65 Gy | 55.6 | 50.0 | 63.2 | 43.8

8. Secondary Outcome: Number of Participants With Severe OM at Varying Cumulative Radiation Doses (Gy)
Description: as for outcome 7
Time Frame: Up to 12 weeks
Population: FAP, 3 participants missing data
Measure: Number; unit: participants
Arm/Group | Placebo | ALD518 (160 mg, OL) | ALD518 (160 mg, R) | ALD518 (320 mg, R)
Number analyzed (Participants) | 24 | 7 | 22 | 20
participants
  35 Gy | 6 | 4 | 6 | 6
  45 Gy | 10 | 5 | 8 | 9
  55 Gy | 12 | 5 | 9 | 11
  65 Gy: number analyzed (Participants) | 18 | 6 | 19 | 16
  65 Gy | 10 | 3 | 12 | 7

9. Secondary Outcome: Duration of Ulcerative and Severe OM
Time Frame: Up to 12 weeks
Population: FAP
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Placebo | ALD518 (160 mg, OL) | ALD518 (160 mg, R) | ALD518 (320 mg, R)
Number analyzed (Participants) | 24 | 7 | 23 | 22
Days
  Ulcerative | 42.0 (23.17) | 55.1 (26.57) | 48.3 (16.71) | 38.0 (29.53)
  Severe | 22.4 (23.28) | 35.1 (28.02) | 22.7 (18.95) | 21.5 (25.01)

10. Secondary Outcome: Time to Onset of Ulcerative and Severe OM
Time Frame: Up to 12 weeks
Population: FAP
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Placebo | ALD518 (160 mg, OL) | ALD518 (160 mg, R) | ALD518 (320 mg, R)
Number analyzed (Participants) | 24 | 7 | 23 | 22
Days
  Ulcerative: number analyzed (Participants) | 22 | 6 | 22 | 18
  Ulcerative | 23.7 (7.05) | 18.7 (5.32) | 22.9 (5.97) | 24.3 (13.37)
  Severe: number analyzed (Participants) | 15 | 5 | 20 | 14
  Severe | 37.0 (11.81) | 26.1 (5.72) | 43.1 (17.55) | 38.0 (15.64)

11. Secondary Outcome: ALD518 Plasma Concentration at Varying Weeks
Time Frame: Baseline and up to 12 weeks
Population: SP
Measure: Mean (Standard Deviation); unit: ug/mL
Arm/Group | ALD518 (160 mg, OL) | ALD518 (160 mg, R) | ALD518 (320 mg, R)
Number analyzed (Participants) | 7 | 23 | 21
ug/mL
  at Baseline: number analyzed (Participants) | 7 | 10 | 9
  at Baseline | 0.0 (0.00) | 0.0 (0.00) | 0.0 (0.00)
  at Week 2: number analyzed (Participants) | 7 | 10 | 8
  at Week 2 | 24.3 (9.98) | 20.6 (3.73) | 32.7 (5.24)
  at Week 4: number analyzed (Participants) | 6 | 10 | 7
  at Week 4 | 18.8 (6.62) | 40.6 (7.53) | 80.6 (20.21)
  at Week 8 (last day of RT): number analyzed (Participants) | 4 | 7 | 6
  at Week 8 (last day of RT) | 31.6 (12.02) | 23.1 (6.64) | 46.9 (13.74)
  at Week 12 (4 weeks post RT): number analyzed (Participants) | 3 | 4 | 2
  at Week 12 (4 weeks post RT) | 16.8 (9.54) | 11.5 (3.10) | 20.6 (14.42)

12. Secondary Outcome: Oral Mucositis Daily Questionnaire (OMDQ) Overall Health Score at Varying Cumulative Radiation Doses (Gy)
Description: Scored on a scale from 0 (worst possible overall health) to 10 (perfect overall health). Higher scores represent better overall health.
Time Frame: Baseline and up to 12 weeks
Population: FAP
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo | ALD518 (160 mg, OL) | ALD518 (160 mg, R) | ALD518 (320 mg, R)
Number analyzed (Participants) | 24 | 7 | 23 | 22
score on a scale
  Baseline: number analyzed (Participants) | 22 | 7 | 20 | 18
  Baseline | 6.5 (1.95) | 8.4 (1.40) | 7.2 (1.66) | 6.7 (2.35)
  35 Gy (up to 12 weeks): number analyzed (Participants) | 24 | 7 | 22 | 20
  35 Gy (up to 12 weeks) | 5.2 (2.08) | 6.6 (2.07) | 5.2 (2.05) | 5.5 (1.91)
  45 Gy (up to 12 weeks): number analyzed (Participants) | 24 | 7 | 21 | 17
  45 Gy (up to 12 weeks) | 5.6 (1.89) | 5.7 (2.14) | 5.4 (1.86) | 5.4 (2.40)
  55 Gy (up to 12 weeks): number analyzed (Participants) | 22 | 7 | 21 | 18
  55 Gy (up to 12 weeks) | 5.1 (1.96) | 5.9 (2.54) | 5.3 (2.22) | 5.1 (2.27)
  65 Gy (up to 12 weeks): number analyzed (Participants) | 18 | 6 | 16 | 14
  65 Gy (up to 12 weeks) | 5.6 (1.79) | 5.7 (3.08) | 5.3 (2.11) | 5.6 (2.37)

13. Secondary Outcome: Functional Assessment of Cancer Therapy - Head and Neck (FACT-HN) Questionnaire Overall Assessment Score at Varying Cumulative Radiation Doses (Gy)
Description: The FACT-HN consists of 28 general + 11 head and neck specific items, each rated on a 0 (not at all) to 4 (very much) Likert type scale. The total score ranges from 0 to 148. Higher scores represent better quality of life.
Time Frame: Baseline and up to 12 weeks
Population: FAP
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo | ALD518 (160 mg, OL) | ALD518 (160 mg, R) | ALD518 (320 mg, R)
Number analyzed (Participants) | 24 | 7 | 23 | 22
score on a scale
  Baseline: number analyzed (Participants) | 22 | 7 | 22 | 20
  Baseline | 116.5 (15.86) | 129.4 (12.63) | 113.8 (19.53) | 111.3 (20.94)
  35 Gy (up to 12 weeks): number analyzed (Participants) | 23 | 7 | 22 | 20
  35 Gy (up to 12 weeks) | 92.9 (20.14) | 100.3 (24.14) | 96.2 (21.18) | 92.2 (19.96)
  45 Gy (up to 12 weeks): number analyzed (Participants) | 24 | 7 | 20 | 19
  45 Gy (up to 12 weeks) | 90.6 (18.18) | 94.7 (30.14) | 89.7 (23.49) | 86.6 (21.34)
  55 Gy (up to 12 weeks): number analyzed (Participants) | 24 | 6 | 19 | 19
  55 Gy (up to 12 weeks) | 89.6 (19.36) | 82.3 (17.79) | 84.4 (25.67) | 81.1 (22.13)
  65 Gy (up to 12 weeks): number analyzed (Participants) | 18 | 6 | 19 | 16
  65 Gy (up to 12 weeks) | 85.2 (18.13) | 93.6 (27.50) | 86.5 (18.00) | 86.5 (23.95)

14. Secondary Outcome: Functional Assessment of Chronic Illness Therapy - Fatigue Questionnaire (FACIT-F) Score at Varying Cumulative Radiation Doses (Gy)
Description: The responses to the 13 items on the FACIT-F questionnaire are each measured on a 5-point Likert scale from 0 (not at all fatigued) to 4 (very much fatigued). The total score ranges from 0 to 52. Higher scores represent less fatigue.
Time Frame: Baseline and up to 12 weeks
Population: FAP
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo | ALD518 (160 mg, OL) | ALD518 (160 mg, R) | ALD518 (320 mg, R)
Number analyzed (Participants) | 24 | 7 | 23 | 22
score on a scale
  Baseline: number analyzed (Participants) | 24 | 7 | 23 | 21
  Baseline | 42.5 (7.26) | 47.6 (3.26) | 42.6 (8.61) | 39.7 (10.94)
  35 Gy (up to 12 weeks): number analyzed (Participants) | 22 | 7 | 22 | 20
  35 Gy (up to 12 weeks) | 31.1 (12.56) | 30.1 (16.63) | 34.0 (9.59) | 31.2 (13.56)
  45 Gy (up to 12 weeks): number analyzed (Participants) | 24 | 7 | 20 | 19
  45 Gy (up to 12 weeks) | 30.3 (11.42) | 28.9 (15.61) | 31.2 (12.33) | 30.4 (11.65)
  55 Gy (up to 12 weeks): number analyzed (Participants) | 24 | 6 | 20 | 19
  55 Gy (up to 12 weeks) | 29.9 (12.95) | 20.8 (14.70) | 28.0 (12.95) | 26.8 (13.71)
  65 Gy (up to 12 weeks): number analyzed (Participants) | 18 | 6 | 19 | 16
  65 Gy (up to 12 weeks) | 29.6 (10.81) | 26.8 (18.71) | 27.3 (9.65) | 29.5 (12.40)

15. Secondary Outcome: Mean Change From Baseline in C-reactive Protein (CRP) Values at Varying Weeks
Description: The level of C-reactive protein (CRP), which can be measured in your blood, increases when there's inflammation in your body.
Time Frame: Baseline and up to 12 weeks
Population: SP. As pre-specified, the two treatment groups that received 160 mg were combined into one 160 mg group for analysis of this endpoint.
Measure: Mean (Full Range); unit: mg/L
Groups:
- ALD518 (160 mg): ALD518 160 mg IV every 4 weeks for a total of 2 doses in open-label (OL) treatment and ALD518 160 mg IV every 3 weeks for a total of 2 doses in randomized (R) treatment
Arm/Group | Placebo | ALD518 (160 mg) | ALD518 (320 mg)
Number analyzed (Participants) | 23 | 32 | 21
mg/L
  Week 1: number analyzed (Participants) | 1 | 3 | 2
  Week 1 | 3.50 [3.5 to 3.5] | -2.20 [-2.4 to -2.1] | -1.15 [-1.7 to -0.6]
  Week 2: number analyzed (Participants) | 22 | 28 | 19
  Week 2 | 8.39 [-13.1 to 73.1] | -6.52 [-31.8 to -0.1] | -14.74 [-75.6 to -0.2]
  Week 3: number analyzed (Participants) | 2 | 4 | 4
  Week 3 | 12.35 [0.8 to 23.9] | -1.75 [-2.3 to -0.4] | -14.78 [-29.2 to -0.6]
  Week 4: number analyzed (Participants) | 20 | 26 | 15
  Week 4 | 4.71 [-12.6 to 38.1] | -6.82 [-31.8 to -0.1] | -14.63 [-75.7 to -0.2]
  Week 5: number analyzed (Participants) | 2 | 3 | 5
  Week 5 | 27.85 [8.6 to 47.1] | -15.50 [-42.2 to -1.9] | -6.30 [-27.7 to -0.6]
  Week 6: number analyzed (Participants) | 16 | 26 | 9
  Week 6 | 20.52 [-9.5 to 98.2] | -6.93 [-31.8 to 0.7] | -11.92 [-75.7 to -0.9]
  Week 8 (last day of RT): number analyzed (Participants) | 17 | 28 | 17
  Week 8 (last day of RT) | 6.51 [-5.3 to 58.8] | -7.84 [-42.8 to -0.1] | -13.96 [-75.7 to -0.2]
  Week 12 (4 weeks post RT): number analyzed (Participants) | 21 | 27 | 16
  Week 12 (4 weeks post RT) | 2.99 [-12.6 to 51.2] | -8.16 [-42.9 to -0.1] | -14.53 [-75.7 to -0.2]

ADVERSE EVENTS:
Time Frame: Up to 15 months for each participant
Description: Safety Population (SP) defined as any subject who received at least 1 dose of ALD518 or placebo. Subjects were analyzed based on the treatment they received. As pre-specified, the two treatment groups that received 160 mg were combined into one 160 mg group.
Arm/Group | Placebo | ALD518 (160 mg) | ALD518 (320 mg)
All-Cause Mortality (participants affected / at risk) | 0/23 | 4/32 | 2/21
Serious Adverse Events (participants affected / at risk) | 7/23 | 15/32 | 8/21
Other Adverse Events (participants affected / at risk) | 22/23 | 32/32 | 21/21
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=23) | ALD518 (160 mg) (N=32) | ALD518 (320 mg) (N=21)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 1
Pancytopenia (Blood and lymphatic system disorders) | 0 | 1 | 0
Acute myocardial infarction (Cardiac disorders) | 0 | 0 | 1
Atrial fibrillation (Cardiac disorders) | 0 | 1 | 0
Coronary artery disease (Cardiac disorders) | 0 | 1 | 0
Myocardial infarction (Cardiac disorders) | 0 | 0 | 1
Tinnitis (Ear and labyrinth disorders) | 0 | 1 | 0
Dysphagia (Gastrointestinal disorders) | 1 | 1 | 0
Nausea (Gastrointestinal disorders) | 0 | 3 | 0
Oral pain (Gastrointestinal disorders) | 1 | 2 | 0
Stomatitis (Gastrointestinal disorders) | 0 | 1 | 0
Tongue haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 1 | 0
General physical health deterioration (General disorders) | 1 | 3 | 0
Pyrexia (General disorders) | 2 | 0 | 0
Abscess limb (Infections and infestations) | 0 | 0 | 1
Bacteraemia (Infections and infestations) | 0 | 1 | 0
Lower respiratory tract infection (Infections and infestations) | 0 | 1 | 0
Pneumonia (Infections and infestations) | 0 | 1 | 1
Pseudomonas infection (Infections and infestations) | 0 | 1 | 0
Accidental overdose (Injury, poisoning and procedural complications) | 0 | 0 | 1
Tracheostomy malfunction (Injury, poisoning and procedural complications) | 0 | 0 | 1
Alanine aminotransferase increased (Investigations) | 0 | 1 | 0
Aspartate aminotransferase increased (Investigations) | 0 | 1 | 0
Blood phosphorous decreased (Investigations) | 0 | 1 | 0
Electrocardiogram ST segment depression (Investigations) | 0 | 1 | 0
Troponin increased (Investigations) | 0 | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 2 | 1 | 1
Tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Cerebrovascular accident (Nervous system disorders) | 0 | 1 | 0
Renal failure acute (Renal and urinary disorders) | 0 | 0 | 1
Renal impairment (Renal and urinary disorders) | 0 | 1 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Obstructive airway disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Pharyngeal haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Tracheal fistula (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=23) | ALD518 (160 mg) (N=32) | ALD518 (320 mg) (N=21)
Anaemia (Blood and lymphatic system disorders) | 4 | 10 | 4
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 0 | 1 | 0
Erythropenia (Blood and lymphatic system disorders) | 1 | 1 | 0
Leukopenia (Blood and lymphatic system disorders) | 7 | 13 | 6
Lymphadenopathy (Blood and lymphatic system disorders) | 1 | 0 | 0
Lymphatic obstruction (Blood and lymphatic system disorders) | 0 | 0 | 1
Lymphopenia (Blood and lymphatic system disorders) | 2 | 3 | 2
Neutropenia (Blood and lymphatic system disorders) | 3 | 10 | 5
Pancytopenia (Blood and lymphatic system disorders) | 0 | 0 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 2 | 9 | 7
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 1
Bundle branch block left (Cardiac disorders) | 0 | 1 | 0
Tachycardia (Cardiac disorders) | 0 | 1 | 1
Deafness (Ear and labyrinth disorders) | 1 | 0 | 0
Ear discomfort (Ear and labyrinth disorders) | 1 | 0 | 1
Ear pain (Ear and labyrinth disorders) | 1 | 5 | 3
Hyperacusis (Ear and labyrinth disorders) | 0 | 1 | 0
Hypoacusis (Ear and labyrinth disorders) | 2 | 2 | 0
Tinnitis (Ear and labyrinth disorders) | 4 | 2 | 2
Vertigo (Ear and labyrinth disorders) | 1 | 1 | 0
Hyperthyroidism (Endocrine disorders) | 0 | 0 | 1
Periorbital oedema (Eye disorders) | 0 | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 3 | 0
Abdominal pain upper (Gastrointestinal disorders) | 2 | 2 | 0
Aphagia (Gastrointestinal disorders) | 2 | 0 | 0
Breath odor (Gastrointestinal disorders) | 0 | 1 | 2
Constipation (Gastrointestinal disorders) | 13 | 22 | 9
Diarrhoea (Gastrointestinal disorders) | 10 | 7 | 3
Dry mouth (Gastrointestinal disorders) | 10 | 11 | 5
Dyspepsia (Gastrointestinal disorders) | 3 | 4 | 1
Dysphagia (Gastrointestinal disorders) | 6 | 12 | 2
Epigastric discomfort (Gastrointestinal disorders) | 0 | 1 | 0
Gastritis (Gastrointestinal disorders) | 0 | 1 | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 | 5 | 2
Glossitis (Gastrointestinal disorders) | 0 | 0 | 1
Glossodynia (Gastrointestinal disorders) | 0 | 1 | 3
Haemorrhoids (Gastrointestinal disorders) | 0 | 0 | 2
Mouth ulceration (Gastrointestinal disorders) | 0 | 1 | 0
Nausea (Gastrointestinal disorders) | 14 | 20 | 14
Odynophagia (Gastrointestinal disorders) | 5 | 5 | 4
Oral mucosal erythema (Gastrointestinal disorders) | 1 | 0 | 0
Oral pain (Gastrointestinal disorders) | 9 | 3 | 7
Regurgitation (Gastrointestinal disorders) | 0 | 1 | 0
Saliva altered (Gastrointestinal disorders) | 1 | 2 | 2
Salivary hypersecretion (Gastrointestinal disorders) | 0 | 1 | 2
Stomatitis (Gastrointestinal disorders) | 2 | 1 | 0
Swollen tongue (Gastrointestinal disorders) | 1 | 0 | 1
Tongue oedema (Gastrointestinal disorders) | 1 | 0 | 0
Tongue ulceration (Gastrointestinal disorders) | 0 | 0 | 2
Vomiting (Gastrointestinal disorders) | 9 | 12 | 10
Asthenia (General disorders) | 3 | 4 | 4
Catheter site haemorrhage (General disorders) | 0 | 0 | 1
Catheter site inflammation (General disorders) | 1 | 0 | 0
Catheter site oedema (General disorders) | 0 | 1 | 0
Catheter site pain (General disorders) | 0 | 1 | 2
Drug intolerance (General disorders) | 0 | 1 | 1
Face oedema (General disorders) | 0 | 1 | 1
Fatigue (General disorders) | 8 | 7 | 5
Hyperthermia (General disorders) | 0 | 1 | 0
Infusion site erythema (General disorders) | 0 | 1 | 0
Local swelling (General disorders) | 0 | 0 | 1
Localized oedema (General disorders) | 0 | 1 | 1
Malaise (General disorders) | 1 | 0 | 0
Oedema peripheral (General disorders) | 1 | 1 | 1
Pyrexia (General disorders) | 2 | 0 | 0
Hyperbilirubinemia (Hepatobiliary disorders) | 0 | 0 | 1
Drug hypersensitivity (Immune system disorders) | 0 | 1 | 0
Bronchitis (Infections and infestations) | 1 | 0 | 0
Diverticulitis (Infections and infestations) | 0 | 1 | 0
Erysipelas (Infections and infestations) | 0 | 0 | 1
Febrile infection (Infections and infestations) | 1 | 0 | 0
Hand-foot-and-mouth disease (Infections and infestations) | 0 | 1 | 0
Herpes simplex (Infections and infestations) | 1 | 0 | 0
Infective glossitis (Infections and infestations) | 0 | 0 | 1
Laryngitis (Infections and infestations) | 0 | 1 | 1
Lower respiratory tract infection (Infections and infestations) | 1 | 0 | 0
Lower respiratory tract infection fungal (Infections and infestations) | 0 | 1 | 0
Nasopharyngitis (Infections and infestations) | 4 | 1 | 3
Oral candidiasis (Infections and infestations) | 11 | 18 | 8
Oropharyngeal candidiasis (Infections and infestations) | 0 | 2 | 0
Pharyngitis (Infections and infestations) | 0 | 1 | 0
Post procedural cellulitis (Infections and infestations) | 1 | 0 | 0
Postoperative wound infection (Infections and infestations) | 1 | 0 | 0
Pseudomonas infection (Infections and infestations) | 1 | 0 | 0
Staphylococcal infection (Infections and infestations) | 0 | 1 | 0
Staphylococcal pharyngitis (Infections and infestations) | 0 | 1 | 0
Tinea cruris (Infections and infestations) | 0 | 1 | 0
Tracheostomy infection (Infections and infestations) | 0 | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 2 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 2 | 0
Viral infection (Infections and infestations) | 0 | 0 | 1
Viral upper respiratory tract infection (Infections and infestations) | 0 | 0 | 1
Accidental overdose (Injury, poisoning and procedural complications) | 0 | 1 | 0
Post procedural haematoma (Injury, poisoning and procedural complications) | 0 | 1 | 0
Post procedural oedema (Injury, poisoning and procedural complications) | 1 | 0 | 1
Radiation fibrosis (Injury, poisoning and procedural complications) | 1 | 0 | 1
Radiation skin injury (Injury, poisoning and procedural complications) | 7 | 8 | 5
Suture related complication (Injury, poisoning and procedural complications) | 0 | 0 | 1
Tracheal obstruction (Injury, poisoning and procedural complications) | 0 | 1 | 0
Alanine aminotransferase increased (Investigations) | 1 | 4 | 1
Aspartate aminotransferase increased (Investigations) | 2 | 2 | 3
Blood alkaline phosphotase increased (Investigations) | 1 | 0 | 1
Blood bicarbonate decreased (Investigations) | 0 | 0 | 1
Blood bilirubin increased (Investigations) | 0 | 1 | 0
Blood calcium decreased (Investigations) | 1 | 0 | 0
Blood chloride decreased (Investigations) | 0 | 1 | 0
Blood cholesterol increased (Investigations) | 0 | 3 | 1
Blood creatinine increased (Investigations) | 1 | 5 | 1
Blood glucose increased (Investigations) | 1 | 0 | 1
Blood potassium decreased (Investigations) | 2 | 0 | 1
Blood pressure diastolic increased (Investigations) | 0 | 1 | 0
Blood pressure increased (Investigations) | 0 | 1 | 0
Blood triglycerides increased (Investigations) | 0 | 2 | 1
Blood urea increased (Investigations) | 1 | 1 | 0
C-reactive protein increased (Investigations) | 1 | 0 | 1
Creatinine renal clearance decreased (Investigations) | 1 | 0 | 0
Electrocardiogram QT prolonged (Investigations) | 0 | 1 | 0
Electrocardiogram change (Investigations) | 1 | 0 | 0
Gamma-glutamyltransferase increased (Investigations) | 0 | 0 | 2
Globulins decreased (Investigations) | 0 | 2 | 1
Haematocrit decreased (Investigations) | 2 | 1 | 2
Haemoglobin decreased (Investigations) | 2 | 3 | 2
Lymphocyte count decreased (Investigations) | 2 | 0 | 2
Mean cell haemoglobin concentration decreased (Investigations) | 1 | 0 | 0
Mean cell haemoglobin decreased (Investigations) | 1 | 0 | 1
Mean cell volume decreased (Investigations) | 1 | 0 | 1
Neutrophil count decreased (Investigations) | 2 | 2 | 6
Platelet count decreased (Investigations) | 2 | 7 | 8
Prealbumin decreased (Investigations) | 0 | 1 | 0
Red blood cell count decreased (Investigations) | 0 | 1 | 1
Renal function test abnormal (Investigations) | 0 | 1 | 0
Reticulocyte count decreased (Investigations) | 0 | 1 | 1
Weight decreased (Investigations) | 7 | 11 | 11
White blood cell count decreased (Investigations) | 2 | 3 | 9
Decreased appetite (Metabolism and nutrition disorders) | 5 | 4 | 1
Dehydration (Metabolism and nutrition disorders) | 1 | 5 | 1
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 0 | 1 | 0
Electrolyte imbalance (Metabolism and nutrition disorders) | 2 | 0 | 0
Gout (Metabolism and nutrition disorders) | 1 | 0 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 2 | 0 | 1
Hypernatraemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Hyperuricaemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Hypocalcaemia (Metabolism and nutrition disorders) | 1 | 2 | 4
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 5 | 4
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 | 2 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 2 | 0 | 1
Hypophagia (Metabolism and nutrition disorders) | 1 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Muscle twitching (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Musculoskeletal discomfort (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 2 | 2 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0
Pain in jaw (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Tumour ulceration (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Ageusia (Nervous system disorders) | 1 | 3 | 2
Aphasia (Nervous system disorders) | 1 | 0 | 0
Aphonia (Nervous system disorders) | 0 | 1 | 0
Cognitive disorder (Nervous system disorders) | 1 | 0 | 0
Dizziness (Nervous system disorders) | 1 | 7 | 1
Drooling (Nervous system disorders) | 1 | 2 | 1
Dysgeusia (Nervous system disorders) | 12 | 11 | 5
Headache (Nervous system disorders) | 8 | 6 | 3
Hypogeusia (Nervous system disorders) | 0 | 0 | 1
Lethargy (Nervous system disorders) | 2 | 0 | 1
Myoclonus (Nervous system disorders) | 0 | 0 | 1
Polyneuropathy (Nervous system disorders) | 1 | 0 | 0
Tongue biting (Nervous system disorders) | 0 | 0 | 1
Tongue paralysis (Nervous system disorders) | 0 | 0 | 1
Agitation (Psychiatric disorders) | 0 | 1 | 1
Anxiety (Psychiatric disorders) | 1 | 4 | 4
Confusional state (Psychiatric disorders) | 0 | 0 | 2
Depressed mood (Psychiatric disorders) | 1 | 0 | 0
Depression (Psychiatric disorders) | 1 | 1 | 0
Drug dependence (Psychiatric disorders) | 0 | 1 | 0
Insomnia (Psychiatric disorders) | 4 | 6 | 1
Chromaturia (Renal and urinary disorders) | 0 | 1 | 0
Nocturia (Renal and urinary disorders) | 0 | 1 | 0
Oliguria (Renal and urinary disorders) | 0 | 1 | 0
Polyuria (Renal and urinary disorders) | 0 | 1 | 0
Proteinuria (Renal and urinary disorders) | 0 | 1 | 0
Renal failure (Renal and urinary disorders) | 1 | 1 | 0
Urinary retention (Renal and urinary disorders) | 0 | 1 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 3 | 7
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 3 | 3 | 3
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 1
Epiglottic oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 4 | 1
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 2
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Increased upper airway secretion (Respiratory, thoracic and mediastinal disorders) | 4 | 4 | 1
Laryngeal oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 4 | 8 | 6
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Sputum discolored (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Sputum increased (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Dermatitis (Skin and subcutaneous tissue disorders) | 3 | 2 | 1
Ecchymosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Erythema (Skin and subcutaneous tissue disorders) | 2 | 2 | 1
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Photodermatosis (Skin and subcutaneous tissue disorders) | 1 | 2 | 1
Pruritis (Skin and subcutaneous tissue disorders) | 0 | 1 | 1
Psoriasis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 0 | 2 | 1
Rash macular (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Rash pruritic (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Skin discoloration (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Skin exfoliation (Skin and subcutaneous tissue disorders) | 1 | 1 | 0
Aortic dilatation (Vascular disorders) | 0 | 0 | 1
Deep vein thrombosis (Vascular disorders) | 0 | 1 | 0
Hypertension (Vascular disorders) | 1 | 2 | 0
Hypotension (Vascular disorders) | 2 | 2 | 2
Lymphoedema (Vascular disorders) | 1 | 1 | 0
Orthostatic hypotension (Vascular disorders) | 0 | 1 | 0
Thrombophlebitis (Vascular disorders) | 1 | 0 | 0
Thrombophlebitis superficial (Vascular disorders) | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No